CLINICAL TRIAL: NCT06814236
Title: Does Patient's Gender Influence 2-way Communication on Anaesthesia Risk Information-Exchange During Informed Consent Obtention? A Prospective Interview-Based Study
Brief Title: Patients Gender Influence on Communication of Anaesthesia Risk
Status: Not yet recruiting | Type: Observational
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Senior Consultant, Sir Ganga Ram Hospital
Other Study IDs: EC/11/24/2618
Record Dates: First submitted 2025-02-01; First posted 2025-02-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anaesthesia Complication
Keywords: gender; anaesthesia risk; informed consent
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males: Patients undergoing elective short-to-moderate duration surgery will be administered a questionnaire based interview at the time of obtaining informed consent
  Interventions: Behavioral: Three-Stage Informed Consent Conversation Model for Anaesthesia Risk profiling
- Females: Patients undergoing elective short-to-moderate duration surgery will be administered a questionnaire based interview at the time of obtaining informed consen
  Interventions: Behavioral: Three-Stage Informed Consent Conversation Model for Anaesthesia Risk profiling

INTERVENTIONS:
Behavioral: Three-Stage Informed Consent Conversation Model for Anaesthesia Risk profiling — Stage 1 Pre-information queries
  Do you know about the risks involved in Anaesthesia?
  If yes, where did you get information about the risks involved with Anaesthesia??
  Which of these do you already know of and what concerns you most?
  Why are you concerned more about that particular risk factor?
  Stage 2 Informing Risks
  The probability or chances of supposed anaesthesia risks could be:
  Probable risk Possible risk Remote risk
  We have the following risk management strategy in place for your reassurance and safety:
  Employing ERAS protocol
  The surgery you are going to undergo, also may have its own set of risks
  Stage 3 Post-information Informing Risks
  In view of the above conversation we had, do you have other point of concern or query on what we have talked about.

SUMMARY:
In Anaesthesia Practice, an Informed consent involves discussing the risks and benefits involved with a certain procedure and its alternatives. Though it is intended to promote patient autonomy and enhance decision-making, the risk profiling, detailing and discussing; generally walks one-way, from the anaesthesiologist to patient/party. This monologue-leaned communication is neither free flowing nor the patients are allowed to 'speak-up-first' on their concerns or queries. Several gaps can be identified including reluctance on the part of the anaesthesiologist to engage the patients in decision making or not upholding the patient preferences; or patient lacking sufficient knowledge to make an informed choice. Therefore, for risk communication, the very context has to be tailored to patient's individual needs.

There is no available study till date which has tried to address as how the communication between patient and the anaesthesiologist is influenced by the 'gender' of the patient concerned. This situates a need to understand how the 'gender' of a patient can influence communication during an Informed consent conversation on anaesthesia risk(s).

The study will explore to decipher if difference(s) in patient's gender influence their perceptions and understanding of anesthesia-related risks, and if the difference will influence the future lines of communication involving either of the gender. This prospective study will be based on conversation model based interview designed to assess the nuances of gender- based differences in risk perception and information exchange during pre-anaesthetic consultations.

DETAILED DESCRIPTION:
The primary goal of informed consent process is to educate patients about their diagnosis, nature and purpose of proposed treatments, potential risks and benefits, available alternatives, and possible outcomes of declining treatment. Though it promotes patient's autonomy, the process also emphasizes their right to decide about their own care, rather than having decisions made solely by the physician. The informed consent framework is built on three essential pillars:

1. Effective risk disclosure by the Clinician (Anaesthesiologist)
2. Patient's perception and understanding of the disclosed risks, including their engagement with the information
3. Patient's ability to evaluate the information, make informed choices, and express a willingness to proceed based on a balanced understanding of the core context and the possible alternatives.

In contemporary medical practice, the informed consent process frequently does not fulfill these criteria. Several gaps have been identified, including, questions about whether anaesthesiologist perceive risk disclosure as a moral obligation or merely a procedural duty, and whether they genuinely respect patient autonomy.

Current evidence indicates that the goal of truly shared decision-making in the context of risk disclosure remains unexplored. The informed consent process often involves an unidirectional flow of information, where the physician discusses the procedure, risks, and potential outcomes with the patient. However, specific risks associated with anaesthesia are frequently under- communicated, as anaesthesiologists' insights into anaesthesia-related complications are not always integrated into pre-operative discussions. For patient-centric care to be administered at par, it is crucial that the risks associated with surgery and anaesthesia are communicated effectively.

The persistence of challenges in risk communication raises several important questions. Research on doctors' perspectives suggests that inadequate communication skills remain a significant barrier, especially when junior doctors or nurses-often tasked with obtaining consent due to the time constraints of senior staff - may not be adequately trained. Unfortunately, in many healthcare settings, the practice remains largely one-sided, with risk information sharing being an informational "dump" rather than a dialogue. These personnel, lacking the specialized knowledge of anaesthesiologists, might not convey the critical information needed for patients to make fully informed decisions.

It is not uncommon that even when patients do engage in discussions, anaesthesiologist, who may assert that the patient lacks sufficient knowledge to make an informed choice, does sometimes not respect their preferences and decisions. This dynamic perpetuates a paternalistic model and undermines the principles of shared decision-making.

The major issue of unidirectional communication, dominated by the healthcare provider, raises the question of whether patients themselves contribute to this imbalance. Some patients may struggle to understand medical information, have limited ability to evaluate risks, forget details quickly, or prefer not to hear about risks due to anxiety. These individuals may adopt a "blunter" coping style, choosing to defer decision-making to the physician and accepting recommendations without seeking detailed explanations. Conversely, "monitor" patients actively seek out information, ask more questions, and may feel dissatisfied if they perceive that the physician has not disclosed all relevant details.

Research has also explored these communication gaps and found that clinicians need to be sensitive to patients' individual needs for information. Patients vary widely in their desire for information based on their educational background, cognitive style, and personal circumstances, etc. Therefore, the study advocates for risk communication to be patient-specific, tailored to meet the distinct informational needs of each individual. Clinicians should assess whether a patient exhibits a "monitor" or "blunter" coping style and adjust their communication strategy accordingly.

Another study highlights the clear role of gender in how patients, particularly women, may agree for surgery even when they feel reluctant or opposed, and despite being hesitant, often sign the consent form due to various factors.

In a study with British women undergoing obstetric and gynecological surgeries, many reported feeling pressured to sign the consent form, pointing to a lack of genuine autonomy. The hospital environment, governed by implicit social norms, creates conditions in which the women felt they had little choice but to comply. This analysis suggests that the informed consent process may not always safeguard patient autonomy and may instead perpetuate a more passive role for patients. This raises broader questions about whether true autonomy in healthcare is realistically attainable and highlights the need for further research on how these dynamics might also affect male patients. However, the study does not mention male patients, suggesting that there may be similar perspectives or vulnerabilities among them that requires exploration.

Despite the existing evidence on gender differences in physician-patient communication, there remain unanswered questions about how these dynamics play out in various medical contexts. There is still a need to understand how gender influences the communication process during the informed consent, particularly in specialties like Clinical Anaesthesia.

A persistent challenge in contemporary Clinical Anaesthesiology practice is the inadequate interaction between patients and anaesthesiologists. This conversation is crucial for respecting patient autonomy, a key principle in Medical Ethics. Despite its importance, risk communication remains inherently challenging, with factors such as varying levels of health literacy, patient anxiety, and provider time limitations influencing its effectiveness. There is not much research on how gender may affect the informed consent obtention, especially in Anaesthesiology practice.

Therefore, further research is desirable to determine whether the observed differences are consistent across diverse clinical settings and how these variations impact patient satisfaction and outcomes during the informed consent process. Additionally, it is essential to explore how the gender of the patients (male and female) may interact to influence communication quality and patient-centered care.

Our study seeks to address this gap by examining whether gender differences influence patients' perceptions and understanding of anaesthesia-related risks. We aim to determine if male and female patients differ in how they interpret, evaluate, or respond to risk information conveyed by a male anaesthesiologist. The study will explore the anaesthesiologist's experience in communicating risk to male versus female patients and whether perceived gender-specific differences towards the information. This proposed investigation will be undertaken using a prospective, interview-based conversation model study designed to assess the nuances of gender-based differences in risk perception during pre-anaesthetic consultations.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients
* Posted for short-2-moderate duration surgery
* Willing to participate
* Education > Bachelors degree
* ASA -I & II physical grade

Exclusion Criteria:

* Patients posted for major surgery
* Patients in for emergency surgery
* ASA III-IV physical grade.
* Patients refusing recording of the interview
* Those looking to their family members to decide upon whether to participate in study • Patients agreeing to recording of the interview but refusing the recorded interview to be evaluated

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing elective surgical procedure under anaesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pre-informed Gender | From beginning of preoperative period to beginning of surgery
  Based on 3-stage informed consent conversation model it will be assessed which gender 'male' or 'female' is pre-informed about anaesthesia concerns and risks when asked

SECONDARY OUTCOMES:
Gender Curosity For Anesthesia Risk Factors | From beginning of preoperative period to beginning of surgery
  Based on 3-stage informed consent conversation model it will be assessed which gender 'male' or 'female' actively engages with the physician for his/her curiosity regarding anaesthesia risk factors not known to them
Gender Perusal for Anaesthesia & Surgical Risk Details | From beginning of preoperative period to beginning of surgery
  Based on 3-stage informed consent conversation model it will be assessed which gender 'male' or 'female' actively seeks to get full details of the probable risk involved in anaesthesia and surgery
Doctor-patient relationship type | From beginning of preoperative period to beginning of surgery
  Based on 3-stage informed consent conversation model it will be assessed what type of doctor-patient relationship (paternalistic, fiduciary, shared decision-making) is established when comparing 'male' and 'female' gender.

CONTACTS AND LOCATIONS:
Overall Officials: Jyotsana Sharma, MSc, Principal Investigator — Sir Ganga Ram Hospital, New Delhi-110060, India; Amitabh Dutta, MD, Study Director — Sir Ganga Ram Hospital, New Delhi-110060, India
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No